CLINICAL TRIAL: NCT01493141
Title: Systemic Effects of Chronic Metal Ion Exposure From Metal-on Metal Hip Resurfacing
Acronym: Metal Ions
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH15402
Record Dates: First submitted 2011-12-07; First posted 2011-12-15 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Osteoarthritis
Keywords: MOMHR; THA; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following markers will be measured using the blood samples:
  1. Serum, erythrocyte, and whole blood cobalt, chromium, and nickel
  2. Serum iron stores:
     Iron, ferritin, transferrin, and total iron binding capacity.
  3. Serum biochemical markers of bone turnover:
     Osteoblast activity markers (including PINP, OC, BALP) Osteoclast activity markers (including NTX-I, CTX-I, ICTP)
  4. Hypothalamo-pituitary axis hormones (in the following order of priority):
     Prolactin LH/FSH + testosterone/oestradiol Growth hormone + IGF-I TSH + Free T3 ACTH + cortisol
  5. Renal function:
     Urea, electrolytes, and creatinine
  6. Hepatic function Liver function tests Clotting screen
  7. Serum lipid profile, full blood count
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MOMHR: Patients who have had metal-on metal hip resurfacing (MOMHR)
- THA: Patients who have had metal-on-polyethylene or ceramic total hip arthroplasty (THA)

SUMMARY:
In recent years hip resurfacing has become a very popular alternative treatment to total hip replacement for the treatment of hip arthritis. This procedure has become particularly common in the young patient with arthritis because of perceived benefits in terms of functional outcome. However, it has recently become apparent that hip resurfacing is associated with a range of adverse events, not typically seen in patients with conventional hip replacement. These include hip fracture, and failure of bone to grow onto the fixation surfaces of the implant. It has also become apparent that hip resurfacing results in the release of high concentrations of dissolved metals in the bloodstream, such as cobalt and chromium. Whilst small concentrations of these metals are essential for normal body functions, such as making red blood cells, in high concentrations their effects can be toxic to many cells and organs of the body, such as bone, the brain, heart, liver and kidneys, as well as disturbing hormones and blood cholesterol levels. Whilst several studies have documented levels of these metal ions of 440 times normal levels in hip resurfacing patients, there are no studies that have examined whether these levels are having a toxic effect on the various organ systems of the body (with the exception of renal function). In this study we plan to explore whether there are differences in bone mineral density, accumulation of metal ions in the brain, and other solid organs, heart and hormonal function between subjects who have had a hip resurfacing 5 or more years previously compared to an individually matched group of subjects after conventional hip replacement.

DETAILED DESCRIPTION:
This is a cross sectional survey in patients who have had hip resurfacing (MOMHR) and subjects who have received a conventional hip replacement (THA) using a metal on plastic or ceramic bearing. Participants in this study will be identified by orthopaedic surgeons from their operating database. An invitation letter will be sent out to the potential participants with an accompanying information sheet and a reply slip. If there is no response then one further letter will be sent out. Those patients who respond to say that they are interested in taking part in the study will then be telephoned by the study team and screened for inclusion/exclusion criteria. If they are eligible and willing to take part after discussions with the investigator, an appointment will be made for them to attend to give informed consent. Participants will be requested not to eat or drink on the morning that they attend for this visit.

There will be an opportunity at this visit for further discussion and explanation of the study requirements with the Investigator before consent is given.

Once consent has been given, the following procedures will be carried out at this visit (Visit 1):

1. Venous blood will be taken by venepuncture (60 mL, approx 4 tablespoons, will be taken) after which the participant will be able to eat breakfast (which will be provided).
2. A urine based pregnancy test will be used in women of child bearing age to exclude pregnant women
3. Participants will complete the Oxford Hip questionnaire, the EQ5D questionnaire and a record of medical history and concomitant medicines under supervision of the student investigator or an experienced research nurse.
4. Whole body bone mineral density assessments will be made using an Hologic Discovery bone densitometer. This will take approximately 10 minutes in total and will be carried out by an experienced research bone density technician
5. An electrocardiogram and an echocardiogram will be performed by an experienced cardiotechnician and later analysed by a Consultant Cardiologist
6. Participants will be given a container and instructions to collect a 24 hour urine sample. This will be returned at the second visit
7. An appointment will be made for the participant to attend for a second visit to the Royal Hallamshire Hospital.

At visit 2 the following procedures will be carried out:

1. Neuropsychological assessments and questionnaires and visual acuity measurement using a Snellen chart.
2. Magnetic resonance imaging (MRI) of the brain using a 3.0T Phillips Intera MRI scanner.
3. MRI of the liver spleen and kidneys using the 3.0T Phillips Intera MRI scanner. Clinical reports will be prepared for all clinical investigations and normal findings will be related to the patient by letter.

Abnormal findings will be reported to the GP and patient with advice for any action as necessary.

ELIGIBILITY:
Inclusion Criteria:

* MOMHR subjects - 35 Men and women at a minimum of 5 years following unilateral or bilateral MOMHR for primary or secondary OA
* Conventional THA subjects - These subjects will be individually (casebycase) matched with MOMHR subjects for age (±3 years), sex, and year of primary arthroplasty surgery (±2 years).

Exclusion Criteria:

* Known inflammatory arthropathy or metabolic bone disease.
* Use of pharmacological doses of estrogen, progestin, androgen, calcitonin, glucocorticoids, or dietary supplements of calcium or vitamin D within the previous 12 months
* Any previous use of bisphosphonate or fluoride therapy (excluding dental prophylaxis)
* Pregnancy
* Subjects who cannot undergo an MRI scan for medical reasons e.g. those with a cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All potential subjects will be identified from the clinical records and registered databases of Mr Wilkinson and Mr Stockley, who are the clinicians who have been directly responsible for the patients clinical care with respect to their hip arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Difference in whole body bone mineral density measured by DXA between patients with MOMHR compared to conventional hip arthroplasty | >5 years after procedure

SECONDARY OUTCOMES:
Serum and urine biochemical markers of osteoclast and osteoblast activity. | >5 years after procedure
Serum, erythrocyte, and whole blood cobalt and chromium levels, measured by inductively-coupled plasma mass spectrometry (ICP MS) | >5 years after procedure
24 hour urinary excretion of cobalt and chromium, measured by ICP MS | >5 years after procedure
Metal ion deposition in solid organs including the brain, liver and kidneys identified by MRI | >5 years after procedure
Cognitive function and visual acuity | >5 years after procedure
Cardiac function, measured by transthoracic echocardiography and electrocardiogram | >5 years after procedure
Renal function measured by serum creatinine, urinary creatinine clearance, urinary N-acetyl-β-D-glucosaminidase (NAG) and Kidney Injury Molecule-1 (Kim-1) | >5 years after procedure
Hepatic function measured by liver function tests and clotting screen | >5 years after procedure
Endocrine function measured by assessment of hypathalamo-pituitary axis hormones | >5 years after procedure
Serum lipid profile and polycythemia, measured by serum triglycerides, cholesterol, and full blood count | >5 years after procedure
Clinical hip replacement function measured by Oxford hip score and EQ-5D | >5 years after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mark JM Wilkinson, Prof, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom